CLINICAL TRIAL: NCT00298285
Title: ABRIDGE: Low Molecular Weight Heparin in Bridging Patients After Mechanical Valve Replacement. A Pilot Study
Brief Title: ABRIDGE: Low Molecular Weight Heparin in Bridging Patients After Mechanical Valve Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABRIDGE
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2006-01

CONDITIONS: Mechanical Valve Replacement; Warfarin Therapy
Keywords: mechanical valve replacement; warfarin
MeSH Terms: interventions — Enoxaparin

INTERVENTIONS:
Drug: enoxaparin

SUMMARY:
The primary aim is to determine the rate of major bleeding and blood clots when using enoxaparin as a bridge to oral blood thinning medication in patients who have undergone mechanical valve replacement.

DETAILED DESCRIPTION:
Patients who undergo mechanical heart valve replacement are usually placed on long-term oral anticoagulation (blood thinning) medication to prevent blood clots from forming on the mechanical valve. This is started in the hospital with intravenous unfractionated heparin; patients must remain in the hospital while on unfractionated heparin. At the same time, an oral blood thinner is started (warfarin). This process is commonly referred to as "bridging." Once the warfarin reaches the proper level, the intravenous heparin is stopped.

This is a single center, non-randomized pilot study using twice a day enoxaparin injections in place of unfractionated heparin as a bridge to warfarin therapy. A total of approximately 100 patients will be enrolled. Patients will be instructed how to give the enoxaparin injections at home. Blood will be drawn every 1-2 days to monitor warfarin levels. Once discharged, patients will continue to have their blood level checked until warfarin is at the correct level, at which point enoxaparin will be discontinued. All patients who develop signs or symptoms of a stroke or abnormal blood clotting will be asked to return for an echocardiogram. An echocardiogram and 12-lead ECG will be done at approximately 30 days after the start of the study.

Additionally the first 100 consecutive patients who fit the inclusion criteria but do not consent to the enoxaparin strategy will be asked to enter a registry that will monitor their hospital stay and information from their routine 30 day follow-up visit will be collected.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all the following will be considered for enrollment.

1. Male or non-pregnant female (negative pregnancy test is required for women of child bearing potential) ≥ 18 of age who are able to provide informed consent and able to self-administer enoxaparin.
2. Body weight ≥ 45kg and ≤ 150kg.
3. Patients who are post prosthetic mechanical valve surgery and will need oral anticoagulation after discharge from the hospital.

   * One who has undergone valve replacement with mechanical prosthesis in the mitral position.
   * One who has undergone valve replacement with mechanical prosthesis in the aortic position.
   * One who has undergone valve replacement with mechanical prosthesis in the tricuspid position.

Exclusion Criteria:

Patients with any of the following will not be eligible for enrollment in the study:

1. Contraindication or sensitivity to unfractionated heparin/ low molecular weight heparin: history of heparin associated thrombocytopenia, heparin induced thrombocytopenia, or heparin induced thrombotic thrombocytopenia syndrome;
2. History of, or current, cardiogenic shock;
3. Active endocarditis (requiring > 4 weeks of antibiotics);
4. Active bleeding or bleeding diathesis;
5. History of gastrointestinal bleeding and /or endoscopically verified ulcer disease within the last three months;
6. Known proliferative diabetic retinopathy or history of intraocular bleeding;
7. Ischemic stroke in the previous three months or any hemorrhagic stroke, known brain tumor, intracranial aneurysm or intracranial AV malformation;
8. Renal insufficiency (cr clearance < 30 cc/min), cr clearance calculation:

   Women = 0.85 x (140 - age) x body weight (kg) / 72 x serum creat (mg/dl), Men = (140 - age) x body weight (kg) / 72 x serum creat (mg/dl), or patient with a renal transplant;
9. Anemia (Hgb < 8 gm/dl);
10. Thrombocytopenia (platelet count < 100 x 109/L);
11. Liver disease demonstrated by ALT > 144u/L
12. Uncontrolled hypertension (systolic blood pressure >180mmHg or diastolic blood pressure >100mmHg);
13. Life expectancy less than 6 months;
14. Moderate pericardial effusion as diagnosed by echo;
15. Concomitant use of clopidogrel, or cyclooxygenase 1 or 2 inhibitors or use within seven days;

Non- medical exclusion

1. Patients unable or unwilling to provide consent.
2. Patients unable or unwilling to have follow-up echocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Study Completion 2006-10

PRIMARY OUTCOMES:
arterial thromboembolism
major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Allan Klein, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States